CLINICAL TRIAL: NCT07294872
Title: A Study Study of Tumor Infiltrating Lymphocytes Injection (GC101/203 TIL) in Patients With Advanced Solid Tumors
Brief Title: A Study of TIL in Advanced Solid Tumors (CZ)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC101/203-2025-CZ-ST
Record Dates: First submitted 2025-12-04; First posted 2025-12-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm B (Experimental): GC101 TILs will be infused i.v. to patients with advanced solid tumors after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: GC101TIL
- Arm A (Experimental): GC203 TILs will be infused i.v. to patients with advanced solid tumors after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.
  Interventions: Biological: GC101TIL

INTERVENTIONS:
Biological: GC101TIL — A tumor sample is resected from each participant and cultured ex vivo to expand the population of Autologous Tumor Infiltrating Lymphocytes Injection (GC101 TIL). After lymphodepletion, patients are infused GC101 TIL.

SUMMARY:
This study is to investigate the safety and efficacy of tumor infiltrating lymphocyte (TIL) therapy in patients with advanced solid tumors. Autologous TILs and gene-edited TILs are expanded from tumor resections and infused i.v. into the patient after NMA lymphodepletion treatment with hydroxychloroquine(600mg,single-dose) and cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* have one the tumor resection for TILs production and successfully produced；
* Age: 18 years to 75years;
* Histologically diagnosed as solid tumors;
* Expected life-span more than 3 months;
* ECOG score 0-1;
* Test subjects have failed standard treatment regimens, and be willing to receive TIL therapy;
* At least 1 evaluable tumor lesion;

Exclusion Criteria:

* with other malignant tumors, except for the malignancies that have been cured, have been inactive for ≥5 years prior to study inclusion and have a very low risk of recurrence; Non-melanoma skin cancer or malignant lentigo with adequate treatment and no evidence of disease recurrence; Carcinoma in situ with adequate treatment and no evidence of disease recurrence;
* Need glucocorticoid treatment, and daily dose of Prednisone greater than 10mg(or equivalent doses of hormones) or outoimmune diseases requiring immunomodulatory treatment;
* Breathe indoor air in a quiet state, and the oxygen saturation of finger pulse is < 95%;
* Human immunodeficiency virus (HIV) infection or anti-HIV antibody positive, active HBV or HCV infection (HBsAg positive and/or anti-HCV positive), syphilis infection or Treponema pallidum antibody positive;
* Significant cardiovascular anomalies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-05-08 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 month
  To characterize the safety profile of GC101 TIL in patients with pancreatic ductal adenocarcinoma who were failed to standard treatment as assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Disease Control Rate (DCR） | Up to 36 months
  Proportion of patients with response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Duration of Response (DOR) | Up to 36 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Progression-Free Survival (PFS) | Up to 36 months
  The time from TIL infusion until disease progression or death from any cause.
Overall Survival(OS) | Up to 36 months
  The time from TIL infusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Huangming Hong, Principal Investigator — Sichuan Cancer Hospital & Institute, Sichuan Cancer Center
Locations (1):
- Sichuan Cancer Hospital & Institute, Sichuan Cancer Center, Chengdu, China